CLINICAL TRIAL: NCT03357211
Title: Accuracy of Maxillary Repositioning During Orthognathic Surgery: a Prospective Observational Descriptive Study in Annecy Genevois Hospital
Brief Title: Accuracy of Maxillary Repositioning During Orthognathic Surgery
Acronym: POMOCOBS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01-POMOCOBS
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Orthognathic Surgery; Maxillofacial Abnormalities
MeSH Terms: conditions — Maxillofacial Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Orthognathic surgery aims to correct jaw position taking into account esthetic and functional criteria (dental occlusion, lip position, breathing...). These surgeries are planned using clinical, radiological and dental cast data. The result of this planning are occlusal splints. Orthognathic surgery had improved in the last decade with 3 dimensions computerized tomography scan (3D CT-Scan) planning and osteosynthesis implants. However the accuracy of the operative results compared to the planned ones has rarely been measured.

DETAILED DESCRIPTION:
Orthognathic surgery aims to correct jaw position taking into account esthetic and functional criteria (dental occlusion, lip position, breathing...). These surgeries are planned only after the end of the growing period and in association with orthodontics. It is necessary to wait the end of facial growth to expect a stable result especially concerning mandibular. The age limit seems to be around 15 to 16 years old for retromandibular deformities and around 18 years old for premandibular deformities.

These surgeries are planned using clinical, radiological and dental cast data. Occlusal splints are made using all these results; these occlusal splints are used during the orthognathic surgery to maintain bones in the planned position.

Since 1993, a navigation system (Orthopilot™) is used, which allow to track jaw position, in real time, with an accuracy around one millimeter and one degree, during orthognathic surgery. This system is routinely used for condyle repositioning after mandibular sagittal split osteotomies; but it is also useful for maxillary navigation and positioning.

The investigator propose to measure the accuracy of the operative results compared to the planned ones, using the Orthopilot™ system.

ELIGIBILITY:
Inclusion Criteria:

* patients needing orthognathic surgery with mobilization of the maxilla via a Le Fort I osteotomy, alone or associated to a mandibular osteotomy, whatever the indication (poor occlusion, sleep apnea, temporo-mandibular dysfunction...)
* patient over 16 years old
* having not expressed any opposition to the collection of his/her personal data for this study (patient him/herself or holder of parental authority in case of patients younger than 18)

Exclusion Criteria:

* pregnancy
* patients deprived of liberty
* protected adult
* patients needing maxillary disjunction

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients needing orthognathic surgery with monobloc mobilization of the maxilla via a Le Fort I osteotomy alone or associated to a mandibular osteotomy, whatever the indication (malocclusion, sleep apnea, temporomandibular dysfunction...), who are adressed to the principal investigator
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Distribution of the translational and rotational shifts of the maxilla between planning and realization | during the surgery
  Shifts will be quantified by 6 components (3 in rotation and 3 in translation) in a coordinate system given by Orthopilot™ navigation system.
  Accuracy of the surgical technic is evaluated by the distribution of the translational and rotational shifts of the maxilla between planning and realization, taking account conformity (when left/right translation is ≤ 1 mm, top/bottom and back/front translations are < 2 mm, frontal rotation is ≤ 1° and axial and sagittal rotations are ≤ 2°), failure (when left/right, top/bottom and back/front translations are > 2 mm, frontal, axial and sagittal rotations are >4°), and non conformity (every other shifts).

SECONDARY OUTCOMES:
Inter-incisal vector | during the surgery
  The inter-incisal vector (that is square root of the sum of each translation shift squared) is calculated by the statistician. It derived from shifts in millimeter and degree measured during surgery by Orthopilot™ navigation system.

CONTACTS AND LOCATIONS:
Overall Officials: Georges Bettega, MD/PhD, Principal Investigator — CH Annecy Genevois